CLINICAL TRIAL: NCT00689338
Title: Open-Label, Non-Comparative, Study Of Intravenous Anidulafungin, Followed Optionally By Oral Voriconazole Or Fluconazole Therapy, For Treatment Of Documented Candidemia/Invasive Candidiasis In Intensive Care Unit Patient Populations
Brief Title: Anidulafungin Candidemia/Invasive Candidiasis Intensive Care Study
Acronym: ICE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Clinical Trials Disclosure Group, Pfizer, Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A8851019
Record Dates: First submitted 2008-05-29; First posted 2008-06-03 (Estimated); Results first posted 2011-05-17 (Estimated); Last update posted 2011-05-30 (Estimated); Status verified 2011-05

CONDITIONS: Invasive Candidiasis
Keywords: Candida; Candidemia; Systemic Candidiasis; ICU; Intensive Care Unit; Critical Care Unit; Anidulafungin; Ecalta; Eraxis; Fluconazole; Voriconazole
MeSH Terms: conditions — Candidiasis, Invasive; Torulopsis; Candidemia; Systemic candidiasis | interventions — Anidulafungin; Fluconazole; Voriconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment Group (Experimental): Option to treat with oral azole therapy following treatment with anidulafungin
  Interventions: Drug: Anidulafungin; Drug: Fluconazole; Drug: Voriconazole

INTERVENTIONS:
Drug: Anidulafungin — Anidulafungin Intravenous Administration
Drug: Fluconazole — Oral Administration of Fluconazole
Drug: Voriconazole — Oral Administration of Voriconazole

SUMMARY:
To evaluate the efficacy and safety of anidulafungin in the treatment of systemic fungal infections in intensive care and critical care unit patients.

ELIGIBILITY:
Inclusion Criteria:

ICU patients with a diagnosis of documented candidemia or invasive candidiasis and belonging to one or more of the following specific populations:

* Post-abdominal surgery.
* Elderly > 65 years old.
* Renal insufficiency / failure / hemodialysis.
* Solid tumor.
* Solid-organ (liver, kidney, lung, heart) transplant recipients.
* Hepatic insufficiency.
* Neutropenic including hematology oncology patients.

Exclusion Criteria:

Patients with poor venous access that would preclude IV drug delivery or multiple blood draws.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 216 (Actual)
Dates: Start 2008-07; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (52):
- Pfizer Investigational Site, Vienna, Austria
- Belgium (5):
  - Pfizer Investigational Site, Brussels
  - Pfizer Investigational Site, Ghent
  - Pfizer Investigational Site, Leuven
  - Pfizer Investigational Site, Liège
  - Pfizer Investigational Site, Yvoir
- Canada (2):
  - Pfizer Investigational Site, Hamilton, Ontario
  - Pfizer Investigational Site, Québec, Quebec
- Czechia (3):
  - Pfizer Investigational Site, Brno
  - Pfizer Investigational Site, Ostrava
  - Pfizer Investigational Site, Prague
- Denmark (2):
  - Pfizer Investigational Site, Koebenhavn OE
  - Pfizer Investigational Site, Odense C
- France (8):
  - Pfizer Investigational Site, Amiens, France
  - Pfizer Investigational Site, Bordeaux, France
  - Pfizer Investigational Site, Clichy, France
  - Pfizer Investigational Site, Lyon, France
  - Pfizer Investigational Site, Marseille, France
  - Pfizer Investigational Site, Montpellier, France
  - Pfizer Investigational Site, Paris, France
  - Pfizer Investigational Site, Villejuif
- Germany (3):
  - Pfizer Investigational Site, Berlin
  - Pfizer Investigational Site, Freiburg im Breisgau
  - Pfizer Investigational Site, Wuppertal
- Greece (2):
  - Pfizer Investigational Site, Kifissia, Athens
  - Pfizer Investigational Site, Haidari, Attica
- Pfizer Investigational Site, Budapest, Hungary
- Italy (4):
  - Pfizer Investigational Site, Pisa
  - Pfizer Investigational Site, Roma
  - Pfizer Investigational Site, Torino
  - Pfizer Investigational Site, Udine
- Netherlands (2):
  - Pfizer Investigational Site, Ede
  - Pfizer Investigational Site, Rotterdam
- Poland (2):
  - Pfizer Investigational Site, Krakow
  - Pfizer Investigational Site, Lodz
- Portugal (3):
  - Pfizer Investigational Site, Coimbra
  - Pfizer Investigational Site, Lisbon
  - Pfizer Investigational Site, Porto
- Romania (2):
  - Pfizer Investigational Site, Iași, Iaşi
  - Pfizer Investigational Site, Bucharest
- Russia (2):
  - Pfizer Investigational Site, Moscow
  - Pfizer Investigational Site, Saint Petersburg
- Slovakia (2):
  - Pfizer Investigational Site, Bratislava
  - Pfizer Investigational Site, Košice
- Turkey (Türkiye) (3):
  - Pfizer Investigational Site, Görükle, Bursa
  - Pfizer Investigational Site, Ankara
  - Pfizer Investigational Site, Trabzon
- Ukraine (2):
  - Pfizer Investigational Site, Dnipropetrovsk
  - Pfizer Investigational Site, Donetsk
- United Kingdom (3):
  - Pfizer Investigational Site, Leeds, West Yorkshire
  - Pfizer Investigational Site, Liverpool
  - Pfizer Investigational Site, London

REFERENCES:
- [Derived] De Rosa FG, Busca A, Capparella MR, Yan JL, Aram JA. Invasive Candidiasis in Patients with Solid Tumors Treated with Anidulafungin: A Post Hoc Analysis of Efficacy and Safety of Six Pooled Studies. Clin Drug Investig. 2021 Jun;41(6):539-548. doi: 10.1007/s40261-021-01024-7. Epub 2021 Apr 23. PMID 33891293
- [Derived] Sganga G, Wang M, Capparella MR, Tawadrous M, Yan JL, Aram JA, Montravers P. Evaluation of anidulafungin in the treatment of intra-abdominal candidiasis: a pooled analysis of patient-level data from 5 prospective studies. Eur J Clin Microbiol Infect Dis. 2019 Oct;38(10):1849-1856. doi: 10.1007/s10096-019-03617-9. Epub 2019 Jul 6. PMID 31280481
- [Derived] Kontoyiannis DP, Bassetti M, Nucci M, Capparella MR, Yan JL, Aram J, Hogan PA. Anidulafungin for the treatment of candidaemia caused by Candida parapsilosis: Analysis of pooled data from six prospective clinical studies. Mycoses. 2017 Oct;60(10):663-667. doi: 10.1111/myc.12641. Epub 2017 Jun 9. PMID 28597967
- [Derived] Kullberg BJ, Vasquez J, Mootsikapun P, Nucci M, Paiva JA, Garbino J, Yan JL, Aram J, Capparella MR, Conte U, Schlamm H, Swanson R, Herbrecht R. Efficacy of anidulafungin in 539 patients with invasive candidiasis: a patient-level pooled analysis of six clinical trials. J Antimicrob Chemother. 2017 Aug 1;72(8):2368-2377. doi: 10.1093/jac/dkx116. PMID 28459966
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A8851019&StudyName=Anidulafungin%20Candidemia/Invasive%20Candidiasis%20Intensive%20Care%20Study%0A

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Adult specific participants were recruited from intensive care unit (ICU) populations.
Pre-assignment Details: Two-hundred twenty one (221) participants were screened; 5 participants were screen failures who did not receive study medication.
Groups:
- Anidulafungin: Anidulafungin: 200 milligrams (mg) Day 1, 100 mg once daily from Day 2 (minimum of 9 days, maximum of 41 days). After Day 10 option to treat with oral azole therapy (voriconazole or fluconazole) at a dose determined by local clinical practice up to a maximum of 56 days from Day 1.
Period: Overall Study
Arm/Group | Anidulafungin
Started | 216
Completed | 73
Not Completed | 143
Not completed — Death | 65
Not completed — Adverse Event | 13
Not completed — Insufficient Clinical Response | 1
Not completed — Lack of Efficacy | 6
Not completed — Other | 8
Not completed — Did not Meet Entrance Criteria | 27
Not completed — Lost to Follow-up | 5
Not completed — Withdrawal by Subject | 3
Not completed — Protocol Violation | 15

BASELINE CHARACTERISTICS:
Arm/Group | Anidulafungin
Number analyzed (Participants) | 216
Age, Customized [Number; unit: participants]
  <18 years | 0
  18 to 44 years | 27
  45 to 64 years | 89
  ≥ 65 years | 100
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 85
  Male | 131

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Global Treatment Response Success at End of Treatment
Description: Global response based on combination of clinical and microbiological outcomes; success defined as clinical response of cure (resolution of signs and symptoms of Candida infection) or improvement (significant, but incomplete resolution of signs and symptoms of Candida infection) in conjunction with microbiological eradication (follow-up culture negative for Candida species) or presumed eradication (follow-up culture not available and clinical response of success).
Time Frame: End of Treatment (Day 14 to Day 56)
Population: Modified Intent-To-Treat (MITT) analysis set: all participants in the ITT population with confirmed diagnosis of candidemia or invasive candidiasis, documented within 96 hours prior to initiation of study treatment or 48 hours after commencing treatment. N excludes participants with missing or unknown global responses.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Anidulafungin
Number analyzed (Participants) | 154
percentage of participants | 69.5 [61.6 to 76.6]

2. Secondary Outcome: Percentage of Participants With Global Response Success at End of Intravenous Treatment (EOIVT)
Description: as for outcome 1
Time Frame: EOIVT (Day 10 up to Day 42)
Population: MITT; N excludes participants with missing or unknown global responses.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Anidulafungin
Number analyzed (Participants) | 157
percentage of participants | 70.7 [62.9 to 77.7]

3. Secondary Outcome: Percentage of Participants With Global Response Success at 2 Weeks After End of Treatment
Description: as for outcome 1
Time Frame: 2 weeks after End of Treatment (Day 14 + 14 up to Day 56 + 14)
Population: MITT; N excludes participants with missing or unknown global responses.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Anidulafungin
Number analyzed (Participants) | 128
percentage of participants | 60.2 [51.1 to 68.7]

4. Secondary Outcome: Percentage of Participants With Global Response Success 6 Weeks After End of Treatment
Description: as for outcome 1
Time Frame: 6 weeks after End of Treatment (Day 14 + 42 up to Day 56 + 42)
Population: MITT; N excludes participants with missing or unknown global responses.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Anidulafungin
Number analyzed (Participants) | 109
percentage of participants | 50.5 [40.7 to 60.2]

5. Secondary Outcome: Time to First Negative Blood Culture
Description: Negative blood culture defined as first negative culture that was not followed by a positive culture within the next 3 days (or 4 days if negative culture was observed on or after Day 10) from start of study medication until end of intravenous treatment (EOIVT). Time to first negative culture includes the first day of study medication.
Time Frame: Day 1 up to Day 42
Population: MITT. N = participants who received a minimum of 3 days of dosing with anidulafungin, excluding participants who experienced invasive candidiasis either at baseline or while on anidulafungin and participants who did not have a first negative blood culture by EOIVT.
Measure: Mean (95% Confidence Interval); unit: days
Arm/Group | Anidulafungin
Number analyzed (Participants) | 87
days | 3.7 [3.0 to 4.3]

6. Secondary Outcome: Day 90 Survival
Description: Percentage of participants known or assumed to be alive on Day 90.
Time Frame: Day 90
Population: MITT
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Anidulafungin
Number analyzed (Participants) | 170
percentage of participants | 54.1 [46.3 to 61.8]
Statistical Analysis 1: Comparison: Anidulafungin; Kaplan-Meier estimate of survival at Day 90 (survivor function); Test type: Superiority or Other; Kaplan-Meier; estimate of survival = 53.8, 95% CI 2-sided [45.9 to 60.9]

7. Secondary Outcome: Time to Successful Intensive Care Unit (ICU) Discharge
Description: Time from start of study medication to successful ICU discharge (by end of treatment [EOT]), defined as being alive on the day after the EOT visit, not being in the ICU on the day after the EOT visit, and being classed as a global treatment success at EOT.
Time Frame: Day 1 up to Day 56
Population: MITT. N = participants who had a successful ICU discharge.
Measure: Mean (95% Confidence Interval); unit: days
Arm/Group | Anidulafungin
Number analyzed (Participants) | 49
days | 16.2 [13.3 to 19.1]

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Anidulafungin
Serious Adverse Events (participants affected / at risk) | 107/216
Other Adverse Events (participants affected / at risk) | 78/216
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Anidulafungin (N=216)
Anaemia (Blood and lymphatic system disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Atrial fibrillation (Cardiac disorders) | 1
Cardiac arrest (Cardiac disorders) | 10
Cardiac failure (Cardiac disorders) | 5
Cardiac failure acute (Cardiac disorders) | 1
Cardio-respiratory arrest (Cardiac disorders) | 5
Cardiopulmonary failure (Cardiac disorders) | 1
Cardiovascular disorder (Cardiac disorders) | 1
Myocardial infarction (Cardiac disorders) | 1
Tachycardia (Cardiac disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 2
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2
Gastrointestinal obstruction (Gastrointestinal disorders) | 1
Haematemesis (Gastrointestinal disorders) | 1
Ileus paralytic (Gastrointestinal disorders) | 1
Intestinal ischaemia (Gastrointestinal disorders) | 2
Intestinal obstruction (Gastrointestinal disorders) | 1
Pancreatic fistula (Gastrointestinal disorders) | 1
Pancreatic necrosis (Gastrointestinal disorders) | 1
Peritonitis (Gastrointestinal disorders) | 2
Rectal haemorrhage (Gastrointestinal disorders) | 1
Stress ulcer (Gastrointestinal disorders) | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Chills (General disorders) | 1
Death (General disorders) | 1
Disease progression (General disorders) | 1
General physical health deterioration (General disorders) | 1
Infusion related reaction (General disorders) | 1
Multi-organ disorder (General disorders) | 2
Multi-organ failure (General disorders) | 12
Sudden death (General disorders) | 1
Haemobilia (Hepatobiliary disorders) | 1
Hepatic failure (Hepatobiliary disorders) | 1
Hepatic haemorrhage (Hepatobiliary disorders) | 1
Pneumobilia (Hepatobiliary disorders) | 1
Abdominal abscess (Infections and infestations) | 1
Cellulitis (Infections and infestations) | 1
Fungaemia (Infections and infestations) | 1
Lung infection pseudomonal (Infections and infestations) | 1
Nosocomial infection (Infections and infestations) | 1
Pancreas infection (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 3
Post procedural infection (Infections and infestations) | 1
Pseudomonal bacteraemia (Infections and infestations) | 1
Sepsis (Infections and infestations) | 6
Septic embolus (Infections and infestations) | 1
Septic shock (Infections and infestations) | 21
Staphylococcal bacteraemia (Infections and infestations) | 1
Urosepsis (Infections and infestations) | 1
Graft thrombosis (Injury, poisoning and procedural complications) | 1
Procedural complication (Injury, poisoning and procedural complications) | 1
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 1
Wound dehiscence (Injury, poisoning and procedural complications) | 1
Body temperature increased (Investigations) | 1
International normalised ratio increased (Investigations) | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Bone neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Metastasis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Cerebral ischaemia (Nervous system disorders) | 1
Convulsion (Nervous system disorders) | 2
Hemiparesis (Nervous system disorders) | 1
Nervous system disorder (Nervous system disorders) | 1
Neurological symptom (Nervous system disorders) | 1
Polyneuropathy (Nervous system disorders) | 1
Somnolence (Nervous system disorders) | 1
Renal failure (Renal and urinary disorders) | 6
Renal failure acute (Renal and urinary disorders) | 1
Urinary bladder haemorrhage (Renal and urinary disorders) | 1
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 2
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 9
Erythema (Skin and subcutaneous tissue disorders) | 1
Abdominal operation (Surgical and medical procedures) | 5
Amputation revision (Surgical and medical procedures) | 1
Debridement (Surgical and medical procedures) | 1
Circulatory collapse (Vascular disorders) | 2
Haemorrhage (Vascular disorders) | 1
Hypotension (Vascular disorders) | 2
Shock (Vascular disorders) | 1
Shock haemorrhagic (Vascular disorders) | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Anidulafungin (N=216)
Anaemia (Blood and lymphatic system disorders) | 16
Thrombocytopenia (Blood and lymphatic system disorders) | 11
Atrial fibrillation (Cardiac disorders) | 11
Tachycardia (Cardiac disorders) | 11
Diarrhoea (Gastrointestinal disorders) | 20
Nausea (Gastrointestinal disorders) | 12
Pyrexia (General disorders) | 12
Hypertension (Vascular disorders) | 16
Hypotension (Vascular disorders) | 15

LIMITATIONS AND CAVEATS:
In a change to the protocol, time to first negative blood/tissue culture will only concern time to first negative blood culture. Lack of regular tissue sampling meant that analysis of time to first tissue culture could not be meaningfully performed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.